CLINICAL TRIAL: NCT03236181
Title: Chronic Effects of Fats on Satiety and Energy Expenditure
Brief Title: Chronic Effects of Fats on Satiety & Energy Needs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is retiring from Center. Research will not continue with a new PI.
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: GFHNRC509
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Overweight; Obesity
Keywords: Energy Expenditure; Appetite; Satiety
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saturated Fat/SFA (Other): 30 grams saturated fat (SFA) in the form of heavy whipping cream will be provided to subject in a mixed meal shake
  Interventions: Other: SFA
- Monounsaturated Fat/MUFA (Other): 30 grams monounsaturated fat (MUFA) in the form of olive oil will be provided to subject in a mixed meal shake
  Interventions: Other: MUFA
- Polyunsaturated Fat Linoleic/PUFA (Other): 30 grams high linoleic polyunsaturated fat (PUFA) in the form of high linoleic sunflower oil will be provided to subject in a mixed meal shake
  Interventions: Other: PUFA
- Polyunsaturated Fat Omega-3/LCn3 (Other): 30 grams high omega-3 polyunsaturated fat (LCn3) in the form of fish oil will be provided to subject in a mixed meal shake
  Interventions: Other: LCn3

INTERVENTIONS:
Other: SFA — High saturated fatty acid/SFA oil source
  Arms: Saturated Fat/SFA
Other: MUFA — High monounsaturated fatty acid/MUFA oil source
  Arms: Monounsaturated Fat/MUFA
Other: PUFA — High polyunsaturated fatty acid (linoleic)/PUFA oil source
  Arms: Polyunsaturated Fat Linoleic/PUFA
Other: LCn3 — High polyunsaturated fatty acid (omega-3)/LCn3 oil source
  Arms: Polyunsaturated Fat Omega-3/LCn3

SUMMARY:
The purpose of this study is to evaluate the effect of dietary fat on satiety (the experience of fullness between one meal and the next) and energy metabolism over an extended period of time (chronic effects). How dietary fat sources affect satiety, appetite and energy use is unclear. The investigators will use a controlled setting for the studies. They want to know if the source of dietary fat alters satiety, satiety hormones, and energy expenditure responses after consuming different diets.

DETAILED DESCRIPTION:
This work will address the interaction of obesity and dietary fatty acids in regulating satiety and energy metabolism. The primary objective is to determine the effects of chronic intake of dietary fatty acids of varied saturation and chain length on satiety, thermogenesis and energy utilization in healthy individuals. The investigators hypothesize that unsaturated fatty acids will 1) increase satiety and 2) increase energy metabolism and that 3) the fatty acid binding protein polymorphisms are associated with reduced energy expenditure in response to dietary fat intake.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between 25.0-34.9 kg/m2
* free of major diagnosed, untreated medical conditions
* non-smoking or use of other tobacco products, including e-cigarettes
* not taking steroid-based medications
* not planning to or currently attempting to gain or lose weight
* willing to comply with study demands
* low intake of long chain omega-3 fatty acids (<0.10 g/d) or willing to reduce intake for 6 weeks prior to starting the study

Exclusion Criteria:

* diagnosed eating disorders
* diabetes (blood sugar ≥ 126 mg/dl)
* hypertension (systolic > 160 mmHg or diastolic > 100 mmHg)
* diagnosed cardiovascular, pulmonary, skeletal and metabolic diseases
* currently pregnant or planning to become pregnant, or lactating
* taking medications known to affect appetite, blood lipids, body composition, body weight, or food intake (appetite control drugs, steroids, antidepressants)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Acute effect of fat intake on energy expenditure as determined by metabolic rate | Incremental Area Under the Curve (iAUC) of metabolic rate from 0 to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Susan Raatz, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No